CLINICAL TRIAL: NCT05867134
Title: Activity Restrictions After Inguinal Hernia Repair
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Eastern Colorado Health Care System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1610664
Record Dates: First submitted 2023-01-30; First posted 2023-05-19 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Inguinal Hernia
Keywords: hernia, recovery, surgery
MeSH Terms: conditions — Hernia, Inguinal; Hernia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Activity as tolerated (Experimental): Instruction will be a treatment group "return to activity as tolerated/comfortable and stop activity if pain present".
  Interventions: Behavioral: Removal of postoperative lifting restrictions
- Standard Lifting Restrictions (No Intervention): Instructions will be "no lifting greater than 20lbs for 6 weeks for open surgery, 2 weeks for minimally invasive surgery".

INTERVENTIONS:
Behavioral: Removal of postoperative lifting restrictions — Patients will be randomized into one of two groups: a control group told to practice standard of care at Eastern Colorado VA with return to activity precautions (6 weeks for open surgery, 2 weeks for minimally invasive surgery) and a treatment group told to "return to activity as tolerated/comfortable and stop activity if pain present".
  Arms: Activity as tolerated

SUMMARY:
This research is intended to be a pilot study to identify differences in outcomes for varied lifting and physical activity precautions following surgical repair of single-sided inguinal hernias. The researchers hypothesize that when given the autonomy to return to activity at the patient's discretion, convalescence will decrease in comparison to a control group given specific precautions to refrain from lifting and strenuous activity. Specific aims include differences in convalescence and surgical outcomes for each group, i.e. rates of complications, hernia recurrence, physical activity assessments pre and postop, and quality of life outcomes.

DETAILED DESCRIPTION:
This study will evaluate lifting restrictions in the postoperative period after inguinal hernia repair. Patients will be consented to the study via in person and electronic methods. Patients will be asked to answer a questionnaire regarding their current pre-operative activity levels in order to establish a baseline. Patients will undergo surgery according to normal medical recommendations and patient preference. Patients will be randomized into one of two groups: a control group told to practice standard of care at Eastern Colorado VA with return to activity precautions (6 weeks for open surgery, 2 weeks for minimally invasive surgery) and a treatment group told to "return to activity as tolerated/comfortable and stop activity if pain present". Patients will be observed in post-operative clinics and asked clinical questions, as well as questionnaires to assess their surgical experience, when they returned to activity, and overall quality of life. Medical charts will be reviewed in order to compare differences in responses and behaviors between the two groups and these data points will be recorded in a password protected document for data analysis.

This study aims to identify if lengthy recommendations for convalescence after inguinal hernia surgery are necessary and determine the impact of allowing the individual patient to have some autonomy in a recommendation to return to physical activity based on their own comfort level. This study could provide the surgical community with a more structured response after this common surgical procedure, as well as potentially reduce convalescence times for individual patients, leading to less economic burden on the individual and the community with returning to work precautions.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of unilateral inguinal hernia
* Must be undergoing surgery
* Must be able to consent

Exclusion Criteria:

* Bilateral inguinal hernia
* Recurrent inguinal hernia
* Surgery scheduled with additional concomitant procedures

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-01-30 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Physiological parameter- Hernia recurrence | 2 years
  Study participants will be followed for 2 years following hernia surgery to evaluate for hernia recurrence in both study arms. Hernia recurrence would be determined by documentation in medical record by surgical teams.
Physiological parameter- Postoperative Complications | 2 months
  Study participants will be evaluated after 2 months for incidence of postoperative complication due to hernia surgery. This includes seroma, hematoma, bleeding, surgical site infection, and wound dehiscence. This will be obtained from participant medical record as documented by clinical providers, primary care providers, surgery, and emergency medicine.

SECONDARY OUTCOMES:
Questionnaire- Postoperative Activity levels | 6 weeks
  Following surgery, study participants will follow specified activity restrictions (per study arm). At the 6 week mark after surgery, participants will complete a survey asking for quantification of vigorous, moderate, walking and sitting activities. Surveys include description of each activity.

CONTACTS AND LOCATIONS:
Overall Officials: Edward Jones, Principal Investigator — VHAECH
Locations (1):
- Rocky Mountain Regional VA Medical Center, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No